CLINICAL TRIAL: NCT02040987
Title: A Single-Center, Randomized, Double-Blinded, Placebo-Controlled, 4-way Cross-over Study to Assess the Effect of a Single Oral Dose of AZD3293 Administration on QTc Interval Compared to Placebo, Using Open-Label AVELOX (Moxifloxacin) as a Positive Control, in Healthy Male Subjects
Brief Title: AZD3293 Thorough QT Study in Healthy Male Volunteers
Acronym: AZD3293TQT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: D5010C00008
Record Dates: First submitted 2014-01-17; First posted 2014-01-20 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Alzheimer's Disease
Keywords: Thorough QT study
MeSH Terms: conditions — Alzheimer Disease | interventions — lanabecestat; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- AZD3293 dose A (Experimental): AZD3293 therapeutic dose oral solution (low dose)
  Interventions: Drug: AZD3293
- AZD3293 dose B (Experimental): AZD3293 supratherapeutic dose oral solution (high dose)
  Interventions: Drug: AZD3293
- Placebo (Placebo Comparator): Placebo oral solution
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator): Moxifloxacin tablet
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: AZD3293 — AZD3293 oral solution - one single dose (low dose).
  Other Names: beta secretase inhibitor
  Arms: AZD3293 dose A
Drug: AZD3293 — AZD3293 oral solution - one single dose (high dose).
  Arms: AZD3293 dose B
Drug: Placebo — Placebo oral solution - one single dose
  Arms: Placebo
Drug: Moxifloxacin — Moxifloxacin tablet - one single dose
  Arms: Moxifloxacin

SUMMARY:
A thorough QT study of AZD3293

DETAILED DESCRIPTION:
A Single-Center, Randomized, Double-Blinded, Placebo-Controlled, 4-way Cross-over Study to Assess the Effect of a Single Oral Dose of AZD3293 Administration on QTc Interval Compared to Placebo, Using Open-Label AVELOX (moxifloxacin) as a Positive Control, in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed, written and dated informed consent prior to any study-specific procedures
2. Healthy male subjects must be able to understand and be willing to comply with study procedures, restrictions and requirements
3. Healthy male subjects aged 18 to 55 years
4. Body weight ≥ 50 to ≤ 100 kg and body mass index (BMI) ≥19 to ≤30
5. Clinically normal findings on physical examination in relation to age, as judged by the investigator.

Exclusion Criteria:

1. History of any clinically significant disease or disorder which may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study
2. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs
3. History of previous or ongoing psychiatric disease/condition including psychosis, affective disorder, anxiety disorder, borderline state and personality disorder
4. History of neurologic disease, including seizures (with the exception of febrile infantile seizures), recent memory impairment or clinically significant head injury
5. History of psychotic disorder among first degree relatives

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The effect of a single dose of AZD3293 low dose and high dose on the change in time-matched QTcF intervals compared with placebo. | Up to 69 days
  The heart rate corrected QT (QTcF) will be calculated using Fridericia's formula

SECONDARY OUTCOMES:
The effect of a single oral dose of moxifloxacin on the changes in time-matched QTcF intervals compared with placebo. | Up to 69 days
  The heart rate corrected QT (QTcF) will be calculated using Fridericia's formula.
The safety and tolerability of AZD3293 in healthy male subjects by assessing a panel of adverse events measures | Up to 69 days
  Physical examination, electrocardiogram, pulse and blood pressure, weight and laboratory variables
Plasma concentrations, AUC, Cmax and tmax of single dose AZD3293 and moxifloxacin in healthy male subjects | Up to 69 days
  AUC(0-t): Area under the concentration versus time curve from time 0 to the time of the last quantifiable concentration to be calculated by a combination of linear and logarithmic trapezoidal methods (linear up-log down) Cmax: Maximum observed plasma concentration obtained directly from the concentration vs. time data tmax: Time to reach Cmax following dose, obtained directly from the concentration vs. time data
The effect of AZD3293 on additional electrocardiogram (ECG) variables (heart rate, RR, PR, QRS, QT and QTcB) | Up to 69 days
  RR: The time between corresponding points on 2 consecutive R waves on ECG. PR: ECG interval measured from the onset of the P wave to the onset of the QRS complex. QRS: ECG interval measured from the onset of the QRS complex to the J point. QT: ECG interval measured from the onset of the QRS complex to the offset of the T wave. QTcB: The heart rate corrected QT calculated using Bazett's formula.

OTHER OUTCOMES:
The relationship between plasma concentrations of AZD3293 and changes in QTcF parameters | Up to 69 days
  The heart rate corrected QT (QTcF) will be calculated using Fridericia's formula

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Goldwater, MD, Principal Investigator — Parexel ECPU Baltimore
Locations (1):
- Research Site, Baltimore, Maryland, United States